CLINICAL TRIAL: NCT03670368
Title: An Interpersonal Relationships Intervention for Improving Cardiovascular Health in Youth
Brief Title: Interpersonal Relationships Intervention and Cardiovascular Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); DePaul University (Other); University of Illinois at Chicago (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Edith Chen, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00203223; R01HL136676 (NIH)
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Mentor/Mentee) (Experimental): Youth in the intervention group will participate in one-on-one mentoring sessions (between mentors and mentees) once per week after school. Mentoring sessions will focus on social relationships, coping behaviors, and healthy lifestyles.
  Interventions: Behavioral: Mentoring
- Comparison group - written materials (Active Comparator): Youth in the comparator group will receive written versions of all materials covered in the mentoring sessions.
  Interventions: Behavioral: Comparison group - written materials

INTERVENTIONS:
Behavioral: Mentoring — The intervention will include one-on-one mentoring sessions held after school, focusing on coping, social relationships, and healthy lifestyles.
  Arms: Intervention (Mentor/Mentee)
Behavioral: Comparison group - written materials — Written materials from the mentoring sessions will be provided to those in the comparison group
  Arms: Comparison group - written materials

SUMMARY:
The purpose of this study is to determine whether random assignment to a mentor-mentee relationship is associated with beneficial cardiovascular health effects in both mentors and mentees.

DETAILED DESCRIPTION:
Participants will be undergraduate students randomly assigned to either being in the mentor or comparison group. A second set of participants will be randomly assigned to either being in the mentee or comparison group. These participants will come from Chicago Public School elementary schools. In total, there will be 125 mentors, 125 comparators, 125 mentees, and 125 comparators. Participants will come for a laboratory visit in which cardiovascular health measures will be taken (details below). Visits will occur once at baseline (before the intervention starts), and once post-intervention. There will be a mid-point assessment of questionnaires. Participants in the intervention group will engage in one-on-one mentoring sessions (mentors together with mentees) once a week after school for the school year. Participants in the comparator group will receive written versions of all materials covered in the mentoring sessions.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate students for mentors
* Chicago Public School students for mentees

Exclusion Criteria:

-

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic symptoms | Change in metabolic symptoms from baseline to approximately 1 year later
  Metabolic symptoms per International Diabetes Federation guidelines
Flow-mediated vasodilation | Change in flow-mediated vasodilation from baseline to approximately 1 year later
  Brachial artery diameter change
HOMA-IR | Change in HOMA-IR score from baseline to approximately 1 year later
  Homeostatic Model Assessment of Insulin Resistance

SECONDARY OUTCOMES:
Pro-inflammatory cytokines | Change from baseline to approximately 1 year later
  Standardized and averaged values of pro-inflammatory cytokines + CRP
Stimulated cytokine production | Change from baseline to approximately 1 year later
  Standardized and averaged values of stimulated pro-inflammatory cytokines
Glucocorticoid sensitivity | Change from baseline to approximately 1 year later
  Standardized and averaged values of cytokine production after stimulation plus addition of cortisol

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No